CLINICAL TRIAL: NCT04547036
Title: Changes in Corneal Endothelial Cell Density After Transscleral ab Interno Glaucoma Gel Stent Implantation
Status: Completed | Type: Observational
Sponsor: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Herbert Reitsamer, Prof. Dr. Herbert Reitsamer, Paracelsus Medical University
Other Study IDs: 0010152018
Record Dates: First submitted 2020-09-08; First posted 2020-09-14 (Actual); Results first posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Glaucoma; Endothelial Cell Loss, Corneal
MeSH Terms: conditions — Glaucoma; Corneal Endothelial Cell Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Endothelial cell count measurment
  Interventions: Device: XEN45

INTERVENTIONS:
Device: XEN45 — Up to 140 consecutive patients with preoperatively recorded endothelial cell counts will be summoned to a consecutive endothelial cell count record and measurement of central corneal thickness postoperatively.

SUMMARY:
The objective of this study is to evaluate the change of endothelial cell count after XEN45 in patients with or without cataract operation.

DETAILED DESCRIPTION:
STUDY OBJECTIVE Corneal endothelial cell loss is a known sequela of glaucoma tube shunt implantation. Big tube shunts show a decrease of endothelial cell count postoperatively (-11.5% after Ahmed glaucoma valves and -12.4% after Molteno shunt 2 years postoperatively). The objective of this study is to evaluate the change of endothelial cell count after XEN45 in patients with or without cataract operation.

PATIENT POPULATION In 140 open angle eyes central endothelial cell counts were recorded preoperatively, before the XEN45 implantation was performed in Dept. Ophthalmology at Paracelsus Medical University Salzburg. XEN45s were already performed in the year 2013-2017 (so up to 5 years) in open angle glaucoma eyes in combination with or without cataract operation. In these eyes central endothelial cell count and central corneal thickness was measured preoperatively and documented in patients records.

STUDY DESIGN A prospective, observational, monocentric trial to evaluate the course of endothelial cell density after the XEN implant. The study will take place in the Dept. Ophthalmology at Paracelsus Medical University Salzburg/SALK.

Up to 140 consecutive patients with preoperatively recorded endothelial cell counts will be summoned to a consecutive endothelial cell count record and measurement of central corneal thickness postoperatively. Informed consents will be obtained from patients, who are interested in participating in the study.

Patients will be assessed for endothelial cell density and the position of the XEN45 measured by anterior segment optical coherence tomography. The distance of the XEN45 to cornea, the angle of the tube, and the tube length in the anterior chamber will be recorded with anterior segment optical coherence tomography. Endothelial cell density will be measured on 3 positions: central, superior-nasal (location of XEN45 implantation), infero-temporal (far away for the XEN45 implant).

OUTCOME PARAMETERS The primary endpoint is the change of central endothelial cell density compared to preoperative data.

Secondary objectives are the differences of supero-nasal and infero-temporal endothelial cell density compared to the central endothelial cell density, and pachymetry compared to preoperative data.

EXAMINATION SCHEDULE Subjects will undergo study visits at the following times: preoperative data (2013-2017) out of patient records, postoperative visit in the year 2018-2020 (1-7 years post XEN45 implantation).

CLINICAL PARAMETERS

The following clinical assessments will be performed at the postoperative examination:

1. Endothelial cell count on different locations of the study eye
2. Central corneal thickness
3. Anterior segment optical coherence tomography (to determine the position of the XEN45)
4. Slit lamp examination of the cornea, anterior segment including gonioscopy (to determine the position of the XEN45), and dilated fundus examination
5. Best corrected visual acuity
6. Measurement of IOP
7. Number and frequency of ocular (glaucoma) medications
8. Ocular symptoms and assessment of complications (especially symptoms, which may be a hint for loss of endothelial cell count)
9. Secondary surgical procedures (if applicable including needlings, lasers, cataract operation, bleb revisions, keratoplasty, secondary IOP lowering procedures, other operations)

ELIGIBILITY:
Inclusion Criteria:

1. Open Angle Glaucoma
2. History past XEN45 implantation with or without combined cataract procedure
3. Available preoperative endothelial cell count data not older than 1 year before XEN operation without any operation between the day of data record and XEN45 operation.
4. Age 18 years or older and of legal age of consent
5. Signed written informed consent
6. Availability, willingness, and sufficient cognitive awareness to comply with examination procedures

Exclusion Criteria:

1. Patients with secondary IOP lowering procedures (excluding SLT, needlings, bleb revisions, YAG lasers, Argon lasers) after XEN implantation will be excluded from analysis, because the secondary IOP lowering procedures may influence endothelial cell count itself. Cataract operations without complications are no exclusion criteria, but have to be recorded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 140 consecutive patients with preoperatively recorded endothelial cell counts will be summoned to a consecutive endothelial cell count record and measurement of central corneal thickness postoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. Ophthalmology and Optometry Paracelsus Medical University, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Groups:
- XEN45 Implantation With and Without Combined Cataract Surgery: Patients with history past XEN45 implantation with and without combined cataract surgery and preoperatively recorded baseline central endothelial cell counts were included for the postoperative examination
Period: Overall Study
Arm/Group | XEN45 Implantation With and Without Combined Cataract Surgery
Started | 129; 155 eyes
Completed | 129; 155 eyes
Not Completed | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: Eyes
Units Other Than Participants: Eyes
Groups:
- XEN45 Implantation With and Without Combined Cataract Surgery: Eyes with a history past XEN45 implantation with and without combined cataract surgery and preoperatively recorded baseline central endothelial cell counts were included for the postoperative examination.
Arm/Group | XEN45 Implantation With and Without Combined Cataract Surgery
Number analyzed (Participants) | 129
Number analyzed (Eyes) | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.4 (10.3)
Sex: Female, Male [Count of Units; unit: Eyes]
  Female | 66
  Male | 89
Ethnicity (NIH/OMB) [Count of Units; unit: Eyes]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 155
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Units; unit: Eyes]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 155
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Eyes]
  Austria | 155

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Cell Count Change
Description: The primary endpoint is the change of central endothelial cell density compared to preoperative data.
Time Frame: baseline compared to 1-5 years postoperative
Measure: Median (95% Confidence Interval); unit: % change compared to baseline
Units Other Than Participants: eyes
Arm/Group | Endothelial Cell Count Measurment
Number analyzed (Participants) | 129
Number analyzed (eyes) | 155
% change compared to baseline
  1 year | 2 [-1 to 5]
  2 years | -1 [-3 to 0]
  3 years | 0 [-3 to 2]
  4 years | -4 [-7 to 1]
  5 years | -1 [-7 to 4]

ADVERSE EVENTS:
Time Frame: 3.7 (range 1.6-6.7) years
Description: The investigators classified the adverse events based on the following definitions according to ISO 14155 (2011).
  Adverse Event (AE) Adverse Device Effect (ADE) Device deficiency Serious Adverse Event (SAE) Serious Adverse Device Effect (SADE)
Arm/Group | XEN45 Implantation With and Without Combined Cataract Surgery
All-Cause Mortality (participants affected / at risk) | 0/129
Serious Adverse Events (participants affected / at risk) | 0/129
Other Adverse Events (participants affected / at risk) | 37/129
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XEN45 Implantation With and Without Combined Cataract Surgery (N=129)
Adult Macular degeneration (Eye disorders) | 20
Conjunctival hyperemia (Eye disorders) | 5
Retinal haemorrhage (Eye disorders) | 3 — Minimum one small spot
conreal guttae (Eye disorders) | 2 — all eyes had pre-existing corneal guttae at baseline visit
Conjuncitval emema (Eye disorders) | 2
Cystoid macular edema (Eye disorders) | 2 — underlying causes were partially pre-existing at baseline visit
Conjuncitval hemorhage (Eye disorders) | 1
Epiretinal membrane (Eye disorders) | 2 — partially pre-existing at baseline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT04547036/Prot_SAP_000.pdf